CLINICAL TRIAL: NCT06126341
Title: Prospective Multi-Center Study to Identify Barriers to Cellular Therapies in Patients With Plasma Cell Disorders PROACT PCD
Brief Title: A Study to Identify Barriers to Cellular Therapies for People With Plasma Cell Disorders
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-166
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; BCMA CAR T-cell therapy; HCT; Memorial Sloan Kettering Cancer Center; 23-166
MeSH Terms: conditions — Multiple Myeloma | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Participant Cohort 1: Relapse/refractory multiple myeloma/RRMM patients less than 70 years of age.
  Interventions: Behavioral: Hospital Anxiety and Depression Scale; Behavioral: Duke-UNC Functional Social Support Questionnaire; Behavioral: Distress Thermometer; Behavioral: FACT-BMT; Behavioral: Psychosocial Assessments of Candidates for Transplantation
- Participant Cohort 2: Relapse/refractory multiple myeloma/RRMM patients 70 years of age or greater
  Interventions: Behavioral: Hospital Anxiety and Depression Scale; Behavioral: Duke-UNC Functional Social Support Questionnaire; Behavioral: Distress Thermometer; Behavioral: FACT-BMT; Behavioral: Psychosocial Assessments of Candidates for Transplantation
- Physician Group 1: Primary Myeloma Therapy: Physicians in this group refer for cellular therapy but do not perform the infusions.
  Interventions: Other: Lecture on the role of cellular therapies in relapse/refractory multiple myeloma/RRMM
- Physician Group 2: CAR Enabled: These physicians can order and infuse CAR T cells but not stem cells.
  Interventions: Other: Lecture on the role of cellular therapies in relapse/refractory multiple myeloma/RRMM
- Physician Group 3: HCT and CAR Enabled: These physicians can order and infuse stem cells and CAR T cells

INTERVENTIONS:
Other: Lecture on the role of cellular therapies in relapse/refractory multiple myeloma/RRMM — Physician investigators will review a lecture on the role of cellular therapies in relapse/refractory multiple myeloma/RRMM that discusses current information in regards to available cellular therapies in RRMM and a proposed treatment algorithm.
  Groups: Physician Group 1: Primary Myeloma Therapy; Physician Group 2: CAR Enabled
Behavioral: Hospital Anxiety and Depression Scale — Depression and anxiety will be assessed using the Hospital Anxiety and Depression Scale (HADS), a 14-item self-rated questionnaire
  Other Names: HADS
  Groups: Participant Cohort 1; Participant Cohort 2
Behavioral: Duke-UNC Functional Social Support Questionnaire — A 14-item, self-administered, multidimensional, functional social support questionnaire has been reduced to an 11 items to a brief and easy-to-complete two-scale, eight-item functional social support instrument.
  Groups: Participant Cohort 1; Participant Cohort 2
Behavioral: Distress Thermometer — The Distress Thermometer is a single-item visual analog scale used to screen cancer patients for the presence of psychological distress
  Other Names: DT
  Groups: Participant Cohort 1; Participant Cohort 2
Behavioral: FACT-BMT — The FACT-BMT Version 4.0 is a 37 item self-report questionnaire that measures the effect of cancer on Quality of Life domains
  Groups: Participant Cohort 1; Participant Cohort 2
Behavioral: Psychosocial Assessments of Candidates for Transplantation — The PACT scale is a single page 10-item rating scale with high inter-rater reliability that has been used extensively in solid organ transplantation
  Other Names: PACT
  Groups: Participant Cohort 1; Participant Cohort 2

SUMMARY:
This is an observational study that will include both participants with relapsed/refractory Multiple Myeloma and their doctors. The purpose of this study is to gather information about the use of hematopoietic cell transplantation/HCT and B-cell maturation antigen /BCMS targeted chimeric antigen receptor/CAR autologous T-cell therapy.

ELIGIBILITY:
Inclusion Criteria:

Patient

* Diagnosis of Multiple Myeloma after January 1, 2017.
* Karnofsky Performance Status > 70%
* ≥ 2 lines of prior therapy
* Anticipated to start new a line of therapy for RRMM within the next 12 months
* Age 18-80 years of age.
* English or Spanish speaking.
* Willing to provide informed consent
* Willing to perform study procedures.

Physician Investigator

* Be a Co-Investigator
* Agree to comply with study procedures

Exclusion Criteria:

Patient

* Active CNS disease
* Patients who already have a definitive plan are to be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering (MSK). If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential participants contacted by their treating physician will be referred to the investigator/research staff of the study. The principal investigator may also screen the medical records of patients with whom they do not have a treatment relationship for the limited purpose of identifying patients who would be eligible to enroll in the study and to record appropriate contact information in order to approach these patients regarding the possibility of enrolling in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2029-05-03 (Estimated); Study Completion 2029-05-03 (Estimated)

PRIMARY OUTCOMES:
Rates of referral | Up to 76 months
  To prospectively estimate the rates of referral and utilization of salvage autologous hematopoietic cell transplantation (HCT) and B cell maturation antigen (BCMA) Targeted Chimeric Antigen Receptor (CAR) autologous T cell therapies among patients with RRMM.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Hartford Healthcare Alliance, Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org